CLINICAL TRIAL: NCT04753242
Title: Psychosocial Care During the COVID-19 Pandemic in Acute Hospitals - an International Online Survey of Psychosomatic, Psychiatric and Psychological Consultation and Liaison (C&L) Services
Brief Title: Psychosocial Care During the COVID-19 Pandemic in Acute Hospitals
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: Req-2020-00861; th21Schaefert
Record Dates: First submitted 2021-02-11; First posted 2021-02-15 (Actual); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Covid-19; COVID-19 Related Psychosocial Burden
Keywords: COVID-19 related psychosocial burden in patients, relatives and staff
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Online survey questionnaire — Self-developed questionnaire based on relevant literature, own experience and consultation with participating professional societies. The survey contains 25 questions on structural and process variables regarding psychosocial care structures that psychosocial C&L services have established in acute hospitals in the context of the COVID-19 pandemic, the implementation and use of COVID-19-related services for patients, relatives and staff, special challenges, as well as needs and wishes for the future. Thereby the survey is aiming at the creation of a data basis for improving the structural and process quality of psychosocial care services through psychosocial C&L services in the context of pandemics, especially the COVID-19 pandemic.

SUMMARY:
Heads of all psychosomatic, psychiatric and psychological consultation and liaison (C&L) services in acute care hospitals across all participating countries will be contacted and asked to participate in this international cross-sectional online survey. The survey consists of questions about care structures and their utilisation that psychosomatic, psychiatric and psychological C&L services have established in acute hospitals in the context of the COVID 19 pandemic.

DETAILED DESCRIPTION:
Background:

The COVID-19 pandemic raised new challenges in supporting patients, relatives and staff for psychosomatic, psychiatric and psychological C&L services in general hospitals worldwide. It is intended to build upon the experience gained so far in order to be well prepared for the future.

Objectives:

The aims of this international online survey are

1. To summarize the efforts made in psychosocial care in the context of the COVID-19 pandemic.
2. To assess the experiences made with the established services so far.
3. To assess the need for networking, cooperation and support.
4. Improvement of psychosocial care in acute hospitals in the context of pandemics.

Study Design:

This health services research project will be carried out as an observational study in the form of an international cross-sectional online survey.

There will be one survey time point. Study reporting will follow the STROBE Statement (Strengthening the Reporting of Observational Studies in Epidemiology).

Ethic approval:

In all participating countries the respective ethics committees were informed about the survey and it was checked with them, how far and what kind of country-specific vote of an ethics committee was necessary. Written statements, declarations or votes were obtained from all participating countries.

Setting:

The heads of all psychosomatic, psychiatric and psychological C&L services in acute care hospitals across all participating countries are contacted and asked to participate. Contact is made via the respective national professional societies and relevant working and interest groups.

Participants This study is an international online survey with psychosomatic, psychiatric and psychological C&L services from 14 European countries (Austria, Belgium, Finland, Germany, France, Greece, Ireland, Italy, Norway, Poland, Portugal, Spain, Switzerland, United Kingdom) as well as parts of Canada (Quebec and Ontario region) and Iran participating.

Country specific regions:

The national coordinators of the participating country provided lists of specific regions for their respective country following the NUTS logic (Nomenclature of Territorial Units for Statistics; https://en.wikipedia.org/wiki/Nomenclature_of_Territorial_Units_for_Statistics), preferably a NUTS level that leads to 5 - 20 NUTS for each country.

Online survey questionnaire:

Self-developed questionnaire based on relevant literature, own experience and consultation with participating professional societies. The survey contains 25 questions on structural and process variables regarding characterization of the participating C&L services, involvement of the respective hospitals in the physical care of COVID-19 patients, structures / organization of psychosocial care for COVID-19 patients in the participating hospitals, specific psychosocial support for patients, relatives and staff established in the participating hospital in the context of COVID-19, communication - How the different target groups were informed about the COVID-19 related psychosocial support services and offers, burden of the COVID-19 pandemic on the psychosocial C&L teams, needs and wishes for the future.

The study questionnaire was translated by a professional company from German into English, French and Italian. Language harmonization and cultural adaptation followed a modified committee-based approach informed by the European Social Survey (ESS) Round 9 Translation Guidelines. Participants are free to choose the language version to be worked on.

ELIGIBILITY:
Inclusion Criteria:

* heads of all psychosomatic, psychiatric and psychological C&L services in acute care hospitals across all participating countries

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The heads of all psychosomatic, psychiatric and psychological C&L services in acute care hospitals across all participating countries will be contacted and asked to participate. Contact will be made via the respective national professional societies and relevant working and interest groups
Sampling Method: Non-Probability Sample
Enrollment: 230 (Actual)
Dates: Start 2020-12-08 (Actual); Primary Completion 2021-10-03 (Actual); Study Completion 2021-10-03 (Actual)

PRIMARY OUTCOMES:
Structural and process quality of COVID-19 related psychosocial C&L services | 6 months
  Data basis for improving quality of COVID-19 related psychosocial C&L services:
  1. characterization of participating C&L services
  2. involvement of respective hospitals in the physical care of COVID-19 patients
  3. structures/ organization of psychosocial care for COVID-19 patients in participating hospitals
  4. specific psychosocial support established in participating hospitals in context of COVID-19 for
     1. patients
     2. relatives
     3. staff
  5. communication strategies - How the different target groups were informed about COVID-19 related psychosocial support services and offers
  6. burden of COVID-19 pandemic on psychosocial C&L teams
  7. needs and wishes of the participating psychosocial C&L services
     1. for support or exchange of experience regarding psychosocial care in the COVID 19 context
     2. for changes / improvements considered essential for the future with regard to psychosocial care services in the participating hospitals in the COVID-19 context

CONTACTS AND LOCATIONS:
Overall Officials: Rainer Schaefert, Prof. Dr. med., Principal Investigator — University Hospital, Basel, Switzerland
Locations (22):
- Medical University of Graz, University Hospital Graz, Graz, Styria, Austria
- Ghent University Hospital, Department of Psychiatry, Ghent, Belgium
- Canada (2):
  - University of Montreal, Department of Psychosomatic Medicine, Montreal
  - TorontoSinai Health, University of Toronto, Department of Psychiatry, Toronto
- Oulu University Hospital and University of Oulu, Oulu, Finland
- Université de Paris, Service de Psychiatrie de l'adulte, Paris, France
- Germany (2):
  - Nuremberg Hospital, Department of Psychosomatic Medicine and Psychotherapy, Nuremberg, Bavaria
  - University Hospital Cologne, Department of Psychosomatics and Psychotherapy, Cologne, North Rhine-Westphalia
- Aristotle University Thessaloniki, Thessaloniki, Greece
- University of Medical Sciences, Department of Psychiatry, Tehran, Iran
- University College Dublin, Dublin, Ireland
- Italy (2):
  - Bologna University, Bologna
  - University of Modena & Reggio Emilia, Modena
- Oslo University Hospital, Oslo, Norway
- Wroclaw Medical University, Wroclaw, Poland
- Portugal (2):
  - Hospital de Santa Maria, Lisbon
  - Universidade Católica Portuguesa Lisboa, Lisbon
- Barcelona University, Barcelona, Spain
- Switzerland (2):
  - University Hospital Basel, Department of Psychosomatic Medicine, Basel, Canton of Basel-City
  - University of Basel, Department of Psychiatry (UPK), Basel
- United Kingdom (2):
  - University of Exeter, Exeter
  - University of York, York

REFERENCES:
- [Derived] van der Feltz-Cornelis CM, Sweetman J, Lee W, Doherty AM, Dineen P, Meinlschmidt G, Vitinius F, Fazekas C, Huber CG, Schaefert R, Stein B. Determinants of workload-related clinician stress levels in general hospital consultation liaison psychiatry services during the COVID-19 pandemic in England and Ireland. Short report. J Psychosom Res. 2024 Feb;177:111584. doi: 10.1016/j.jpsychores.2023.111584. Epub 2023 Dec 30. PMID 38181547
- [Derived] Schaefert R, Stein B, Meinlschmidt G, Roemmel N, Huber CG, Hepp U, Saillant S, Fazekas C, Vitinius F. COVID-19-Related Psychosocial Care in General Hospitals: Results of an Online Survey of Psychosomatic, Psychiatric, and Psychological Consultation and Liaison Services in Germany, Austria, and Switzerland. Front Psychiatry. 2022 Jun 24;13:870984. doi: 10.3389/fpsyt.2022.870984. eCollection 2022. PMID 35815043